CLINICAL TRIAL: NCT05557513
Title: Evaluating the Effectiveness and Feasibility of Community Based SARS-CoV-2 Antigen Rapid Diagnostic Testing (Ag-RDT) in the Myanmar Migrant Community, Tak Province Along the Thai Myanmar Border for Controlling Coronavirus Transmission
Brief Title: Research on Community Based ATK Test Study to Control Spread of COVID-19 in Migrant Community
Acronym: CATK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VIR22002
Record Dates: First submitted 2022-06-15; First posted 2022-09-28 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19; Thailand; ATK; SARS-CoV-2 antigen rapid diagnostic testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: For primary objective (Ag-RDT (arm 1) and no Ag-RDT (arm 2)) 74 clusters (37 in each arm) Approximate 5,500 participants in arm 1 and 5,500 participants in arm 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ag-RDT (arm 1) (Active Comparator): Symptomatic /suspected COVID-19 participant or close contact/family members of COVID-19 patient will be tested with Ag RDT and also involve in awareness-raising campaign with mask distribution.
  Interventions: Device: STANDARD Q COVID-19 Ag Test
- No Ag-RDT (arm 2) (No Intervention): No community based Ag RDT testing but there has routine ATK or RT-PCR test by Thai health authorities if local health volunteer finds symptomatic or suspected COVID-19 or close contact with positive cases in their villages. The participant also involves in awareness-raising campaign with mask distribution.

INTERVENTIONS:
Device: STANDARD Q COVID-19 Ag Test — Device Name: STANDARD Q COVID-19 Ag Test Manufactured by SD Biosensor, Inc., Korea
  Purpose: To detect COVID-19 (Its manufacture specification sensitivity was at 84.97% and specificity 98.4%)
  Arms: Ag-RDT (arm 1)

SUMMARY:
Thousands of migrants from Myanmar have arrived in Thailand for their safety, better living standards and employment opportunities. They are often in Thailand illegally and have poor access to the Thai health care system. This underutilization not only puts their health at risk but may also put the general public's health at risk. During the COVID-19 pandemic, migrants often have no access to diagnostic tests even though global health actors are focused on accelerating access to COVID-19 testing. SARS-CoV-2 testing is one of the most effective and necessary means of mitigating the COVID-19 pandemic.

The overarching goal of this study is to provide evidence on effectiveness and feasibility of community-based SARS-CoV-2 antigen rapid diagnostic test (Ag-RDT) application in the Myanmar migrant community, Tak Province along the Thai Myanmar border as part of test-trace-isolation strategies to fight COVID-19.

After the study has been completed, the study team will have evidence to inform policymakers on whether community based SARS-CoV-2 Ag-RDT test-trace-isolate strategy is effective and feasible to fight COVID-19 where there is limited or no access to COVID-19 testing in the Myanmar migrant communities.

DETAILED DESCRIPTION:
This study plan to recruit people who are living in the Maramat and Pohphra Myanmar migrant community or returning to community from outside.

This study includes seroprevalence survey (secondary objective) at the beginning and at the post-intervention of study to estimate the percentage of people in a population who have antibodies against SARS-CoV-2 by capillary blood collection from finger prick. This secondary objective will be achieved through a substudy. In the substudy, 427 participants will be studied from 7 clusters that will be randomly sampled from the parent study for the Ag RDT arm and similarly 427 participants will be studied from 7 clusters that will be randomly sampled from the parent study for the No Ag RDT arm. There will be two cross-sectional surveys in each of these two arms one at baseline and the other at post-intervention. The aim will be to compare the post-intervention percentage of people in a population who have antibodies against SARS-CoV-2 by capillary blood collection from finger prick between the two arms.

The two arms of the substudy will be managed as follows:

One arm (Arm 1): Symptomatic /suspected COVID-19 participant or close contact/family members of COVID-19 patient will be tested with Ag RDT and also involve in awareness-raising campaign with mask distribution.

One arm (Arm 2): No community based Ag RDT testing but there has routine ATK or RT-PCR test by Thai health authorities if local health volunteer finds symptomatic or suspected COVID-19 or close contact with positive cases in their villages. The participant also involves in awareness-raising campaign with mask distribution.

Ten focus group discussion (FGD) with community members will be conducted to find out the attitudes and perception of community members on the use of community based SAR COV2 Ag-RDTs testing in Myanmar migrant community for prevention control of COVID-19 in the study area.

The overarching goal of this study is to provide evidence on effectiveness and feasibility of community-based SARS-CoV-2 antigen rapid diagnostic test (Ag-RDT) application in the Myanmar migrant community, Tak Province along the Thai Myanmar border for test-trace-isolation strategies to fight COVID-19.

After the study has been completed, depending upon the study finding, study team believe that study team can propose to policymakers to recognize the effectiveness and feasibility of community-based SARS-CoV-2 Ag-RDT's test-trace-isolate strategies to fight COVID-19 where there is limited or no access to COVID-19 testing in the Myanmar migrant communities

This study was funded by The Foundation for Innovative New Diagnostics (FIND). The grant reference number is U-22008

ELIGIBILITY:
1. For Ag RDT arm (primary objective)

   1. Inclusion Criteria

      * *Symptomatic COVID-19 patient/suspected COVID-19 or **close contact/family members of COVID-19 patient
      * Participant at any age living in chosen clusters of Maramat and Pohphra Myanmar migrant community
      * Participant or parent/guardian/caretaker is willing and able to give informed consent for participation in the study.
   2. Exclusion Criteria

      * Known history of a COVID-19 positive test result within the last 21 days
2. For No Ag RDT arm (primary objective)

   1. Inclusion Criteria

      * Participant at any age living in chosen cluster of Maramat and Pohphra Myanmar migrant community
      * Symptomatic COVID-19 patient/suspected COVID-19 or **close contact/family members of COVID-19 patient who agrees to go for routine Thai COVID-19 ATK or RT-PCR test
      * Participant or parent/guardian/caretaker is willing and able to give informed consent for participation in the study
   2. Exclusion Criteria

      * Not living in chosen clusters in Maramat and Pohphra Myanmar migrant community

   note: *Symptomatic or suspected COVID-19: Acute onset of ANY THREE OR MORE of the following signs or symptoms: Fever, cough, general weakness/fatigue1, headache, myalgia, sore throat, coryza, dyspnoea, anorexia/nausea/vomiting1, diarrhoea, altered mental status (1 Signs separated with slash (/) are to be counted as one sign) Reference: WHO-2019-nCoV-Surveillance_Case_Definition-2020.2-eng (5).pdf

   note: **1 Person who stayed close to or had conversation with COVID-19 patient(s) for >5 minutes, or was exposed to the patient's cough or sneeze; 2 Individual who stayed in enclosed spaces with poor ventilation together with COVID-19 patient(s) for >30 minutes, for instance, in air-conditioned bus, commuter vane, or air-conditioned room; Reference: g_HCWs_3Mar22.pdf (moph.go.th)
3. For seroprevalence survey (secondary objective)

   1. Inclusion Criteria

      * Participant at any age living in chosen clusters of Maramat and Pohphra Myanmar migrant community
      * Participant or parent/guardian/caretaker is willing and able to give informed consent for participation in the study.
   2. Exclusion Criteria

      * Refusal to give informed consent, or contraindication to venepuncture
4. For Focus group discussion (FGD)

   1. Inclusion Criteria

      * Age 18 years and above
      * Living in chosen clusters of Maramat and Pohphra migrant communities
      * Participant is willing and able to give informed consent for participation in the study.
   2. Exclusion Criteria

      * Not living in chosen clusters of Maramat and Pohphra migrant communities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1310 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the differences in number of cases detected per 1,000 people between the Ag-RDT and No Ag-RDT intervention arms. | through study completion, an average of 3 months
  The number of cases per 1,000 will be estimated and summarised per group/arm and will compared between groups

SECONDARY OUTCOMES:
Compare the seroprevalence of SAR COV2 antibody between Ag-RDT Arm (1) and No Ag-RDT Arm (2) | through study completion, an average of 3 months
  Seroprevalence of SAR COV2 antibody in each of the groups at baseline and at post-intervention surveys.
Find out about the attitudes of community members on the use of community based SAR COV2 Ag-RDTs testing in Myanmar migrant community | through study completion, an average of 3 months
  Attitudes of community participants towards community base SAR COV2 Ag-RDTs use.
Find out about the perception of community members on the use of community based SAR COV2 Ag-RDTs testing in Myanmar migrant community | through study completion, an average of 3 months
  Perception of community participants towards community base SAR COV2 Ag-RDTs use.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Thaw Htwe MIn, Principal Investigator — Shoklo Malaria Research Unit (SMRU) 69/30 Ban Tung Road, Maesot63110, Tak, Thailand Tel: +66-087-307-0971
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of MORU, will be de-identified and may be shared in fully anonymised form with other researchers in accordance with the current Data Sharing Policy. (https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs ).
Time Frame: For data and records will be retained for five years following completion of the study. Afterwards, all the identifiable data from source documents as well as the electronic database will be destroyed. De-identified data will be archived in SMRU for the purpose of pooled or secondary data analysis.
  Data may be used alone or in combination with data from related studies in secondary analyses. Any data published in the peer-reviewed medical literature will protect the identity of the participant.
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs